CLINICAL TRIAL: NCT05549700
Title: The Fascicular Anatomy of Nerve May Influence the Muscular Activity of the Biceps Femoris After Applying Ultrasound-guided Percutaneous Neuromodulation
Brief Title: The Application of Neuromodulation in Sciatic Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Sciatic nerve and NMP
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Healthy
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common fibular nerve group (Experimental): The subjects of this group will receive electric nerve stimulation on the sciatic nerve through a lateral approach to stimulate the behavior corresponding to the common fibular nerve
  Interventions: Other: Neuromodulation
- Tibial nerve group (Experimental): The subjects of this group will receive electric nerve stimulation on the sciatic nerve through a lateral approach to stimulate the behavior corresponding to the tibial nerve
  Interventions: Other: Neuromodulation

INTERVENTIONS:
Other: Neuromodulation — Ultrasound-guided percutaneous neuromodulation will be applied. The protocol used was 5 seconds of stimulation, 55 seconds of rest for 5 minutes at a frequency of 100 Hz and a phase duration of 350 microseconds

SUMMARY:
The objective of this study will be to analyze the muscle activity of the short head (SHBF) and long head of the biceps femoris (LHBF) after the application of ultrasound-guided percutaneous neuromodulation (NMP) in the tibial or common fibular nerve compartment of the sciatic nerve.

Authors will recruit healthy subjects and they will receive asymmetric biphasic rectangular current through a needle into the sciatic nerve. The sample was divided into two groups: one to which the technique was applied in the lateral compartment and another group, in the medial compartment of the nerve. The protocol used was 5 seconds of stimulation, 55 seconds of rest for 5 minutes at a frequency of 100 Hz and a phase duration of 350 microseconds. The electrical activity (recruitment of muscle fibers and maximum contraction) of the SHBF and LHBF and the muscle strength of the knee flexors were recorded by requesting the participants isometric flexion of the knee in the prone position. The percentage of change of each variable was also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Subjects that have lumbar area of the back, scoliosis, lower limb dysmetria
* Subjects undergone any surgical intervention in the lumbar area or lower limbs
* Subjects that present acute or unresolved injury in the last 6 months in the lower limbs
* Subjects under treatment drug treatment
* Subjects that they are afraid of needles or electric current
* Subjects with epileptic
* Pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Electrical muscular activity | 3 months
  recruitment of muscle fibers, measured by electromyography (microvolts)
muscle strength of the knee flexors | 3 months
  strength measured by dynamometer (Kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Blanca, Seville, Sevile, Spain

REFERENCES:
- [Derived] Paez-Rodriguez J, Olivo-Ruiz I, Romero-Morales C, De-la-Cruz-Torres B. The fascicular anatomy of the sciatic nerve may not influence the muscular activity of the biceps femoris after applying percutaneous electrical nerve stimulation: a randomized clinical trial. Acupunct Med. 2024 Dec;42(6):326-333. doi: 10.1177/09645284241300176. Epub 2024 Nov 21. PMID 39569806